CLINICAL TRIAL: NCT04968912
Title: A Randomized, Placebo-controlled, Double-blind, Multicenter Study to Assess the Efficacy and Safety of Nipocalimab in Adults With Primary Sjogren's Syndrome (pSS)
Brief Title: A Study of Nipocalimab in Adults With Primary Sjogren's Syndrome (pSS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CR109062; 80202135SJS2001 (Other: Janssen Research & Development, LLC); 2021-000665-32 (EudraCT Number)
Expanded Access: NCT05221619 (Temporarily not available)
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Placebo (Placebo Comparator): Participants will receive placebo intravenously (IV) every 2 weeks (q2w) through Week 22 along with standard of care treatments ([including ophthalmic drops, artificial tears and saliva, punctum plugs, and secretagogues], and/or one immunomodulator with or without low-dose glucocorticosteroids).
  Interventions: Other: Placebo; Drug: Standard of Care Treatment
- Group 2: Nipocalimab Dose 1 (Experimental): Participants will receive nipocalimab dose 1 IV q2w through Week 22 along with standard of care treatments ([including ophthalmic drops, artificial tears and saliva, punctum plugs, and secretagogues], and/or one immunomodulator with or without low-dose glucocorticosteroids).
  Interventions: Drug: Nipocalimab; Drug: Standard of Care Treatment
- Group 3: Nipocalimab Dose 2 (Experimental): Participants will receive nipocalimab dose 2 IV q2w through Week 22 along with standard of care treatments ([including ophthalmic drops, artificial tears and saliva, punctum plugs, and secretagogues], and/or one immunomodulator with or without low-dose glucocorticosteroids).
  Interventions: Drug: Nipocalimab; Drug: Standard of Care Treatment

INTERVENTIONS:
Other: Placebo — Placebo infusion will be administered intravenously.
  Arms: Group 1: Placebo
Drug: Nipocalimab — Nipocalimab dose 1 and dose 2 infusions will be administered intravenously.
  Other Names: JNJ-80202135; M281
  Arms: Group 2: Nipocalimab Dose 1; Group 3: Nipocalimab Dose 2
Drug: Standard of Care Treatment — Standard of care treatment including ophthalmic drops, artificial tears and saliva, punctum plugs, and secretagogues, and/or one immunomodulator with or without low-dose glucocorticosteroids will be administered topically/orally.

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of nipocalimab in participants with primary Sjogren's syndrome (pSS) versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Meets classification criteria for primary Sjogren's syndrome (pSS) by the 2016 American College of Rheumatology (ACR) / European League Against Rheumatism (EULAR) at the time of screening (results either obtained during screening or documented in the participant's medical history are acceptable to fulfill these criteria for Schirmer's test, unstimulated salivary flow test, ocular staining score, or labial salivary gland biopsy), and was diagnosed with pSS no less than 26 weeks prior to screening
* At screening is seropositive for antibodies to pSS-associated antigen A (Ro/Sjogren's syndrome-related antigen A [SSA])
* Total Clinical European League Against Rheumatism Sjogren's Syndrome Disease Activity Index (clinESSDAI) score greater than or equal to (>=) 6
* At least one abnormal laboratory marker of pSS-related inflammatory disease activity, and at least low activity in one or more specified European League Against Rheumatism Sjogren's Syndrome Disease Activity Index (ESSDAI) domains
* It is recommended to be up to date on all age-appropriate vaccinations prior to screening per routine local medical guidelines. It is strongly recommended that participants will have completed a locally-approved (or emergency use-authorized) coronavirus disease 2019 (COVID-19) vaccination regimen at least 2 weeks prior to study related visits or procedures. Study participants should, follow applicable local vaccine labelling, guidelines, and standards-of-care for participants receiving immune-targeted therapy will be followed when determining an appropriate interval between vaccination and study enrollment

Exclusion Criteria:

* Has any confirmed or suspected clinical immunodeficiency syndrome not related to treatment of his/her pSS or has a family history of congenital or hereditary immunodeficiency unless confirmed absent in the participant
* Comorbidities (for example, asthma, chronic obstructive pulmonary disease) which have required 3 or more courses of systemic glucocorticoids within the previous 12 months
* Has any unstable or progressive manifestation of pSS that is likely to warrant escalation in therapy beyond permitted background medications and/or has severely active pSS
* Has received oral cyclophosphamide within 3 months or intravenous (IV) cyclophosphamide within 6 months prior to first administration of study intervention
* Has Sjogren's syndrome overlap syndromes where another confirmed autoimmune rheumatic or systemic inflammatory condition (for example, rheumatoid arthritis [RA], systemic lupus erythematosus [SLE], scleroderma, inflammatory bowel disease [IBD]) is the primary diagnosis or has clinical manifestations that, in the opinion of the investigator, or the sponsor or sponsor's representative, are likely to interfere with the investigator's ability to assess pSS manifestations

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Clinical European League Against Rheumatism Sjogren's Syndrome Disease Activity Index (clinESSDAI) Score at Week 24 | Baseline to Week 24
  The clinESSDAI is a validated tool used in clinical studies to measure the systemic disease activity in participants with primary Sjogren's syndrome. The clinESSDAI includes 11 domains divided into 3-4 activity levels, where zero represents no activity and low, medium, and high scores can vary in numerical value depending on the domain.

SECONDARY OUTCOMES:
Change from Baseline in European League Against Rheumatism (EULAR) Sjogren Syndrome Patient Reported Index (ESSPRI) Score at Week 24 | Baseline to Week 24
  The ESSPRI is a patient-reported assessment of the severity of dryness, fatigue, and pain associated with primary Sjogren's Syndrome. Participants are asked to rate the severity of dryness, fatigue and pain over the past 2 weeks on a numeric rating scale (NRS), ranging from 0 "no symptoms (dryness, fatigue or pain)" to 10 "maximal imaginable (dryness, fatigue, pain)". A global score, calculated as the mean of the 3 domain scores, ranges from 0 to 10, with higher scores reflecting greater (worse) symptom severity.
Improvement of Greater than or Equal to (>=) 4 Points from Baseline in ESSDAI Score (Minimal Clinically Important Improvement) at Week 24 | Baseline to Week 24
  The ESSDAI is a validated tool used in clinical studies to measure the systemic disease activity in participants with primary Sjogren's syndrome. The ESSDAI includes 11 to 12 domains divided into 3-4 activity levels, where zero represents no activity and low, medium, and high scores can vary in numerical value depending on the domain.
Improvement of >= 4 Points from Baseline in clinESSDAI Score (Minimal Clinically Important Improvement) at Week 24 | Baseline to Week 24
  The clinESSDAI is a validated tool used in clinical studies to measure the systemic disease activity in participants with Sjogren's syndrome. A minimal clinically important improvement in clinESSDAI is defined as a decrease of at least 4 points in the composite clinESSDAI score.
ESSPRI Response at Week 24 | Week 24
  ESSPRI response defined as a decrease of one point or a decrease of >= 15 percent (%) from baseline (minimal clinically important improvement) at Week 24 will be reported.
Disease Response as Assessed by Sjögren's Tool for Assessing Response (STAR) Composite Score at Week 24 | Week 24
  Disease response by STAR of >= 5 at Week 24 will be reported. STAR is a composite tool that incorporates measures of disease activity (clinESSDAI), symptoms (ESSPRI), glandular function and systemic disease activity biomarkers to assess disease activity.
Improvement in Disease Activity Level by >= 1 Level in at Least One clinESSDAI or ESSDAI Domain at Week 24 | Week 24
  Improvement in disease activity level by >= 1 level in at least one clinESSDAI or ESSDAI domain (biological, hematological, cutaneous, constitutional, lymphadenopathy and lymphoma, and glandular) at Week 24 will be reported.
Improvement from Baseline in >= 3 of 5 Composite of Relevant Endpoints for Sjogren's Syndrome (CRESS) Categories at Week 24 | Baseline to Week 24
  Improvement from baseline in >= 3 of 5 CRESS categories at week 24 will be reported. CRESS is a composite tool that incorporates measures of disease activity (clinESSDAI), symptoms (ESSPRI), glandular function and systemic inflammation to assess disease activity.
Percentage of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to 30 weeks
  An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Percentage of Participants with Adverse Events of Special interests (AESIs) | Up to 36 weeks
  Percentage of participants with AESIs will be reported. Treatment-emergent adverse events associated with the following situations are considered as AESIs: severe infections, severe hypoalbuminemia or hypogammaglobulinemia.
Percentage of Participants with Treatment-emergent Serious Adverse Events (SAEs) | Up to 30 weeks
  Treatment-emergent SAEs are defined as SAEs with onset or worsening on or after date of first dose of study treatment.
Percentage of Participants with TEAEs Leading to Treatment Discontinuation | Up to 30 weeks
  Percentage of participants with TEAEs leading to treatment discontinuation will be reported. TEAEs are defined as AEs with onset or worsening on or after date of first dose of study treatment.
Percentage of Participants with Clinically Significant Abnormalities in Vital Signs | Up to 36 weeks
  Percentage of participants with clinically significant abnormalities in vital signs (including temperature, pulse/heart rate, respiratory rate, and blood pressure) through end of study visit will be reported.
Percentage of Participants with Clinically Significant Abnormalities in Laboratory Parameters | Up to 36 weeks
  Percentage of participants with clinically significant abnormalities in laboratory parameters (including hematology, blood chemistry, urinalysis, and blood coagulation) through end of study visit will be reported.
Serum Concentration of Nipocalimab Over Time | Up to Week 30
  Serum concentrations of nipocalimab over time in participants receiving active study intervention will be reported.
Number of Participants with Antibodies to Nipocalimab (Anti-drug Antibodies [ADAs] and Neutralizing Antibodies [NAbs]) | Up to Week 36
  Number of participants with antibodies to nipocalimab (ADAs and NAbs) in participants receiving active study intervention will be reported.
Number of Participants with Change from Baseline in Biomarkers | Baseline to Week 36
  Number of participants with change from baseline in biomarkers (C-reactive protein [CRP], erythrocyte, total immunoglobulin [Ig]G, IgG1, IgG2, IgG3, IgG4) will be reported.
Number of Participants with Change from Baseline in Autoantibodies | Baseline to Week 36
  Number of participants with change from baseline in autoantibodies (anti-Sjogren's syndrome related antigen A (anti-Ro/SSA), anti-Sjogren's syndrome related antigen B (anti-La/SSB), rheumatoid factor [RF] and antinuclear antibody [ANA]) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (69):
- United States (25):
  - Anniston Medical Clinic, Anniston, Alabama
  - Arizona Arthritis and Rheumatology Research PLLC, Glendale, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Mesa, Arizona
  - St. Jude Heritage Medical Group, Fullerton, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - Colorado Arthritis Associates, Denver, Colorado
  - Denver Arthritis Clinic, Denver, Colorado
  - Rheumatology Associates Of South Florida, Boca Raton, Florida
  - Bay Area Arthritis and Osteoporosis, Brandon, Florida
  - Centre for Rheumatology, Immunology and Arthritis, Fort Lauderdale, Florida
  - University of Florida Health Jacksonville, Jacksonville, Florida
  - Omega Research Consultants, Orlando, Florida
  - Clinical Investigation Specialists, Gurnee, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - St. Paul Rheumatology P A, Eagan, Minnesota
  - North Mississippi Medical Clinics, Tupelo, Mississippi
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Columbia Arthritis Center, Columbia, South Carolina
  - West Tennessee Research Institute, Jackson, Tennessee
  - Dr. Ramesh Gupta, Memphis, Tennessee
  - Austin Regional Clinic, Austin, Texas
  - Trinity Clinical Research, LLC, Carrollton, Texas
- France (5):
  - CHU de Grenoble Hopital Albert Michallon, La Tronche
  - Centre Hospitalier Le Mans, Le Mans
  - Hopital Saint Joseph, Marseille
  - Hopital Pitie Salpetriere, Paris
  - CHRU Hôpital de Hautepierre, Strasbourg
- Germany (6):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Uniklinik Köln, Cologne
  - Universitatsklinikum Carl Gustav Carus Dresden, Dresden
  - Hamburger Rheuma Forschungszentrum II, Hamburg
  - medius KLINIK KIRCHHEIM, Kirchheim unter Teck
  - Universitatsklinikum Tubingen, Tübingen
- Italy (5):
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia Presidio Spedali Civili, Brescia
  - P.O. Vittorio Emanuele Azienda Ospedaliero Universitaria 'Policlinico Vittorio Emanuele', Catania
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Japan (6):
  - Tokyo Metropolitan Tama Medical Center, Fuchū
  - Nagasaki University Hospital, Nagasaki
  - Hokkaido University Hospital, Sapporo
  - St. Luke's International Hospital, Tokyo
  - Nihon University Itabashi Hospital, Tokyo
  - University of Tsukuba Hospital, Tsukuba
- Netherlands (2):
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Erasmus Medisch Centrum, Rotterdam
- Poland (10):
  - Nasz Lekarz Przychodnie Medyczne, Bydgoszcz
  - Szpital Uniwersytecki nr 2 im dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Zespolu Opieki Zdrowotnej w Konskich, Gmina Końskie
  - Malopolskie Badania Kliniczne Sp z o o, Krakow
  - REUMED Zespol Poradni Specjalistycznych Filia nr 2, Lublin
  - Centrum Medyczne, Poznan
  - Medycyna Kliniczna, Warsaw
  - Narodowy Instytut Geriatrii Reumatologii i Rehabilitacji im prof dr hab med Eleonory Reicher, Warsaw
  - Centrum Medyczne AMED Targowek, Warsaw
  - Centrum Medyczne Oporow, Wroclaw
- Portugal (2):
  - Instituto Portugues de Reumatologia, Lisbon
  - ULSAM, EPE - Hospital Conde de Bertiandos, Ponte de Lima
- Spain (6):
  - Hosp Univ A Coruna, A Coruña
  - Hosp Reina Sofia, Córdoba
  - Hosp. de Merida, Mérida
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Infanta Luisa, Seville
- Taiwan (2):
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency

REFERENCES:
- [Derived] Noaiseh G, Sivils KL, Campbell K, Idokogi J, Lo KH, Liva SG, Leu JH, Dhatt H, Ma K, Leonardo S, Li H, Hubbard JJ, Gottenberg JE. Efficacy and safety of nipocalimab in patients with moderate-to-severe Sjogren's disease (DAHLIAS): a randomised, phase 2, placebo-controlled, double-blind trial. Lancet. 2025 Nov 22;406(10518):2435-2448. doi: 10.1016/S0140-6736(25)01430-8. Epub 2025 Oct 24. PMID 41284548